CLINICAL TRIAL: NCT00863304
Title: A PHASE 3 RANDOMIZED, DOUBLE BLIND PLACEBO AND NAPROXEN CONTROLLED MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE HIP OR KNEE
Brief Title: Tanezumab in Osteoarthritis of the Hip or Knee (2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091018
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis
Keywords: monoclonal antibody RN624 PF-04383119 nerve growth factor anti-nerve growth factor OA pain arthritis
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: tanezumab 10 mg
- 2 (Experimental)
  Interventions: Biological: tanezumab 5 mg
- 3 (Active Comparator)
  Interventions: Drug: naproxen
- 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: tanezumab 10 mg — tanezumab 10 mg one dose at weeks 0 and 8
  Arms: 1
Biological: tanezumab 5 mg — tanezumab 5 mg one dose at weeks 0 and 8
  Arms: 2
Drug: naproxen — naproxen 1000 mg daily for 16 weeks
  Arms: 3
Other: placebo — placebo to match tanezumab and naproxen dosing
  Arms: 4

SUMMARY:
Test the efficacy and safety of 2 doses of tanezumab compared with naproxen and placebo in patients with osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the hip or knee according to Kellgren-Lawrence x-ray grade of 2

Exclusion Criteria:

* pregnancy or intent to become pregnant
* BMI greater than 39
* other severe pain, significant cardiac, neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2009-06-09 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (95):
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - Saadat Ansari, MD, Huntsville, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Clinical Research Advantage, Inc. / Central Arizona Medical Associates, PC, Mesa, Arizona
  - Novara Clinical Research, Mesa, Arizona
  - Clinical Research Advantage, Inc., Mesa, Arizona
  - Central Phoenix Medical - Clinical Research Advantage, Phoenix, Arizona
  - Paradigm Clinical, Inc, Tucson, Arizona
  - eStudySite, Chula Vista, California
  - Orthopedic Physicians of Colorado, PC, Englewood, California
  - University Parks Hematology/Oncology, Englewood, California
  - Edinger Medical Group and Research Center, Fountain Valley, California
  - Valley Research, Fresno, California
  - Lakewood Orthopedic Medical & Surgical Group, Lakewood, California
  - High Desert Medical Group Research for Life, Lancaster, California
  - Premiere Clinical Research, LLC, Long Beach, California
  - Miracle Mile Medical Center, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Del Carmen Medical Center, Reseda, California
  - Probe Clinical Research, Corp., Santa Ana, California
  - Lawrence P.McAdam, MD, A Medical Corporation, Thousand Oaks, California
  - Westlake Medical Center, Westlake Village, California
  - Peak Anesthesia and Pain Management, Centennial, Colorado
  - Denver Internal Medicine Group, Denver, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Colorado Hematology, Englewood, Colorado
  - Colorado Orthopedic Consultants, PC, Englewood, Colorado
  - American Clinical Research, LLC, Englewood, Colorado
  - Norwalk Medical Group, Norwalk, Connecticut
  - Rheumatology Consultants of Delaware, Lewes, Delaware
  - HeartCare, Bradenton, Florida
  - In Vivo Clinical Research, Inc, Doral, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Kendall South Medical Center, Inc, Miami, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - HeartCare Research, Sarasota, Florida
  - Tampa Medical Group PA, Tampa, Florida
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Pasadena Pharmacy, Lexington, Kentucky
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - L-Marc Research Center, Louisville, Kentucky
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Miray Medical Center, Brockton, Massachusetts
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - Planters Clinic, Port Gibson, Mississippi
  - St. John's Medical Research Institute, Inc., Springfield, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Diagnositc Center of Medicine, Henderson, Nevada
  - Independent Clinical Researchers, Las Vegas, Nevada
  - Wolfson Medical Center, Las Vegas, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - Medex Healthcare Research, Inc., New York, New York
  - SPRI Bronx LLC, The Bronx, New York
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Orthopedic & Sports Medicine Consultants, Middletown, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Physicians' Research, Inc, Zanesville, Ohio
  - PrimeCare of Southeastern Ohio, Inc, Zanesville, Ohio
  - Cor Clinical Research, LLC, Oklahoma City, Oklahoma
  - The Family Healthcare Center, PA, Clinton, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Low Country Rheumatology, PA, North Charleston, South Carolina
  - The Carolina Center for Rheumatology and Arthritis Care, PA, Rock Hill, South Carolina
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - South Austin Orthopedics, Austin, Texas
  - Tekton Research Inc. - Research Office, Austin, Texas
  - Texas Orthopedic Specialists, Grapevine, Texas
  - Foundation for Southwest Orthopedic Research, Houston, Texas
  - Southwest Orthopedic Group, Houston, Texas
  - The Neurology Center, Houston, Texas
  - Gill Orthopedic Center, Lubbock, Texas
  - Robert R. King, M.D., PA, Lubbock, Texas
  - AZ Clinical Research, Sugar Land, Texas
  - Spring Clinical Research, Sugar Land, Texas
  - Sugar Land Med-Ped, P.A., Sugar Land, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Incorporated/Foothill Family Clinic South, Salt Lake City, Utah
  - Commonwealth Orthopedics & Rehabilitation , P.C., Arlington, Virginia
  - IntegraTrials, LLC, Arlington, Virginia
  - Virginia Hospital Center, Arlington, Virginia
  - HypotheTest, LLC, Roanoke, Virginia
  - Empirical Clinical Trials, LLC, Selah, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Ekman EF, Gimbel JS, Bello AE, Smith MD, Keller DS, Annis KM, Brown MT, West CR, Verburg KM. Efficacy and safety of intravenous tanezumab for the symptomatic treatment of osteoarthritis: 2 randomized controlled trials versus naproxen. J Rheumatol. 2014 Nov;41(11):2249-59. doi: 10.3899/jrheum.131294. Epub 2014 Oct 1. PMID 25274899
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091018&StudyName=Tanezumab%20in%20osteoarthritis%20of%20the%20hip%20or%20knee%20%282%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to tanezumab (PF-04383119) intravenous (IV) infusion over 5 minutes at Baseline (Day 1) and Week 8 along with placebo matched to naproxen tablet orally twice daily at Baseline (Day 1), and at Weeks 4, 8 and 12.
- Tanezumab 5 mg + Placebo: Participants received tanezumab (PF-04383119) 5 milligram (mg) IV infusion over 5 minutes at Baseline (Day 1) and Week 8 along with placebo matched to naproxen tablet orally twice daily from Baseline up to Week 12.
- Tanezumab 10 mg + Placebo: Participants received tanezumab (PF-04383119) 10 mg IV infusion over 5 minutes at Baseline (Day 1) and Week 8 along with placebo matched to naproxen tablet orally twice daily from Baseline up to Week 12.
- Naproxen + Placebo: Participants received naproxen 500 mg tablet orally twice daily at Baseline (Day 1), Weeks 4, 8 and 12 along with placebo matched to tanezumab (PF-04383119) IV infusion at Baseline (Day 1) and Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Started | 212 | 212 | 213 | 212
Treated | 209 | 211 | 209 | 211
Completed | 18 | 27 | 26 | 21
Not Completed | 194 | 185 | 187 | 191
Not completed — Adverse Event | 10 | 4 | 14 | 16
Not completed — Lost to Follow-up | 1 | 5 | 4 | 2
Not completed — Lack of Efficacy | 57 | 26 | 30 | 28
Not completed — Withdrawal by Subject | 19 | 14 | 20 | 18
Not completed — Other | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 6 | 2 | 0
Not completed — Randomized, but not Treated | 3 | 1 | 4 | 1
Not completed — Entered extension study | 101 | 129 | 113 | 125

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of randomized IV study medication (either tanezumab or placebo IV).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo | Total
Number analyzed (Participants) | 209 | 211 | 209 | 211 | 840
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 6 | 13 | 14 | 14 | 47
  45 to 64 years | 133 | 133 | 134 | 126 | 526
  Greater than or equal to (>=) 65 years | 70 | 65 | 61 | 71 | 267
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 134 | 128 | 136 | 534
  Male | 73 | 77 | 81 | 75 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). BOCF method was used to impute missing values. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.41 (1.38) | 7.27 (1.38) | 7.37 (1.39) | 7.30 (1.41)
  Change at week 16 | -2.14 (2.74) | -3.32 (2.77) | -3.03 (3.05) | -2.61 (2.70)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Analysis of Covariance (ANCOVA) was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; Least Square (LS) Mean Difference = -1.13, 95% CI 2-sided [-1.65 to -0.62], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.80, 95% CI 2-sided [-1.32 to -0.29], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.090, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.45, 95% CI 2-sided [-0.96 to 0.07], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.69, 95% CI 2-sided [-1.21 to -0.17], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.175, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.36, 95% CI 2-sided [-0.87 to 0.16], Standard Error of Mean 0.26

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Week 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Physical function refers to participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated maximum difficulty. Total score range for WOMAC physical function subscale score was 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated worse physical function.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.04 (1.49) | 6.83 (1.56) | 7.09 (1.52) | 6.95 (1.64)
  Change at Week 16 | -1.75 (2.53) | -3.01 (2.64) | -2.86 (2.98) | -2.25 (2.51)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.23, 95% CI 2-sided [-1.71 to -0.75], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.99, 95% CI 2-sided [-1.48 to -0.51], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.067, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.94 to 0.03], Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.77, 95% CI 2-sided [-1.26 to -0.29], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.54, 95% CI 2-sided [-1.03 to -0.05], Standard Error of Mean 0.25

3. Primary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 16: Baseline Observation Carried Forward (BOCF)
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1=very good (no symptom and limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). BOCF method was used to impute missing values. Here, 'overall number of participants' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 3.46 (0.65) | 3.36 (0.56) | 3.40 (0.61) | 3.48 (0.61)
  Change at Week 16 | -0.49 (0.80) | -0.80 (0.89) | -0.80 (1.00) | -0.66 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.34, 95% CI 2-sided [-0.50 to -0.18], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.32, 95% CI 2-sided [-0.48 to -0.16], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.078, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.14, 95% CI 2-sided [-0.30 to 0.02], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.18, 95% CI 2-sided [-0.34 to -0.02], Standard Error of Mean 0.08

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 2, 4, 8, and 12: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Change at Week 2 | -2.11 (2.15) | -2.64 (2.48) | -2.42 (2.64) | -2.92 (2.42)
  Change at Week 4 | -2.29 (2.38) | -3.48 (2.55) | -3.27 (2.82) | -2.98 (2.33)
  Change at Week 8 | -2.23 (2.46) | -3.46 (2.65) | -3.06 (2.81) | -2.85 (2.39)
  Change at Week 12 | -2.12 (2.69) | -3.40 (2.76) | -3.24 (3.02) | -2.78 (2.63)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 2: ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.49, 95% CI 2-sided [-0.94 to -0.05], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.214, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.28, 95% CI 2-sided [-0.73 to 0.16], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.76, 95% CI 2-sided [-1.21 to -0.32], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.234, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.27, 95% CI 2-sided [-0.18 to 0.72], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.48, 95% CI 2-sided [0.04 to 0.93], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 4: ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.16, 95% CI 2-sided [-1.63 to -0.70], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.96, 95% CI 2-sided [-1.42 to -0.49], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.64, 95% CI 2-sided [-1.11 to -0.18], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.52, 95% CI 2-sided [-0.99 to -0.05], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.193, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.31, 95% CI 2-sided [-0.78 to 0.16], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 8: ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.20, 95% CI 2-sided [-1.68 to -0.73], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.80, 95% CI 2-sided [-1.28 to -0.32], Standard Error of Mean 0.24
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.62, 95% CI 2-sided [-1.10 to -0.14], Standard Error of Mean 0.24
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.58, 95% CI 2-sided [-1.06 to -0.10], Standard Error of Mean 0.24
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.464, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.18, 95% CI 2-sided [-0.66 to 0.30], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 12: ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.22, 95% CI 2-sided [-1.72 to -0.72], Standard Error of Mean 0.26
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.04, 95% CI 2-sided [-1.55 to -0.54], Standard Error of Mean 0.26
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.014, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.63, 95% CI 2-sided [-1.14 to -0.13], Standard Error of Mean 0.26
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.023, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.59, 95% CI 2-sided [-1.09 to -0.08], Standard Error of Mean 0.26
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.114, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.92 to 0.10], Standard Error of Mean 0.26

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in Pain Subscale at Weeks 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). LOCF method was used to impute missing values. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.41 (1.38) | 7.27 (1.38) | 7.37 (1.39) | 7.30 (1.41)
  Change at Week 2 | -2.11 (2.15) | -2.64 (2.48) | -2.42 (2.64) | -2.92 (2.42)
  Change at Week 4 | -2.42 (2.36) | -3.57 (2.49) | -3.35 (2.79) | -3.04 (2.35)
  Change at Week 8 | -2.48 (2.39) | -3.59 (2.57) | -3.39 (2.75) | -3.05 (2.39)
  Change at Week 12 | -2.58 (2.63) | -3.79 (2.58) | -3.73 (2.84) | -3.12 (2.56)
  Change at Week 16 | -2.64 (2.67) | -3.80 (2.58) | -3.58 (2.87) | -3.07 (2.66)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.49, 95% CI 2-sided [-0.94 to -0.05], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.214, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.28, 95% CI 2-sided [-0.73 to 0.16], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.76, 95% CI 2-sided [-1.21 to -0.32], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.234, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.27, 95% CI 2-sided [-0.18 to 0.72], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.48, 95% CI 2-sided [0.04 to 0.93], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.13, 95% CI 2-sided [-1.59 to -0.67], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.91, 95% CI 2-sided [-1.37 to -0.45], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.59, 95% CI 2-sided [-1.05 to -0.13], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.023, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.54, 95% CI 2-sided [-1.00 to -0.07], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.175, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.32, 95% CI 2-sided [-0.78 to 0.14], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.09, 95% CI 2-sided [-1.55 to -0.63], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.88, 95% CI 2-sided [-1.34 to -0.41], Standard Error of Mean 0.24
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.56, 95% CI 2-sided [-1.03 to -0.10], Standard Error of Mean 0.24
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.52, 95% CI 2-sided [-0.99 to -0.06], Standard Error of Mean 0.24
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.190, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.31, 95% CI 2-sided [-0.78 to 0.15], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.15, 95% CI 2-sided [-1.63 to -0.68], Standard Error of Mean 0.24
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.07, 95% CI 2-sided [-1.55 to -0.60], Standard Error of Mean 0.24
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.52, 95% CI 2-sided [-0.99 to -0.04], Standard Error of Mean 0.24
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.64, 9% CI 2-sided [-1.12 to -0.16], Standard Error of Mean 0.24
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.023, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.56, 95% CI 2-sided [-1.04 to -0.08], Standard Error of Mean 0.24
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 5 mg + Placebo; Week 16: ANCOVA was performed with treatment as main effects, baseline value, index joint as a covariate, and study site as a random effect; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.12, 95% CI 2-sided [-1.60 to -0.64], Standard Error of Mean 0.24
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.87, 95% CI 2-sided [-1.35 to -0.39], Standard Error of Mean 0.25
Statistical Analysis 23: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.092, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.90 to 0.07], Standard Error of Mean 0.25
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.71, 95% CI 2-sided [-1.19 to -0.23], Standard Error of Mean 0.25
Statistical Analysis 25: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.94 to 0.03], Standard Error of Mean 0.25

6. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.04 (1.49) | 6.83 (1.56) | 7.09 (1.52) | 6.95 (1.64)
  Change at Week 2 | -1.60 (2.12) | -2.34 (2.37) | -2.33 (2.50) | -2.52 (2.40)
  Change at Week 4 | -1.77 (2.24) | -3.04 (2.50) | -2.94 (2.80) | -2.55 (2.36)
  Change at Week 8 | -1.76 (2.31) | -3.00 (2.61) | -2.83 (2.79) | -2.40 (2.29)
  Change at Week 12 | -1.71 (2.49) | -3.06 (2.66) | -2.95 (2.95) | -2.47 (2.45)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.70, 95% CI 2-sided [-1.12 to -0.27], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.66, 95% CI 2-sided [-1.09 to -0.23], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.82, 95% CI 2-sided [-1.25 to -0.39], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.572, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.12, 95% CI 2-sided [-0.31 to 0.55], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.467, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.16, 95% CI 2-sided [-0.27 to 0.59], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.28, 95% CI 2-sided [-1.74 to -0.83], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.12, 95% CI 2-sided [-1.58 to -0.66], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.73, 95% CI 2-sided [-1.19 to -0.27], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.55, 95% CI 2-sided [-1.01 to -0.09], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.101, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.39, 95% CI 2-sided [-0.85 to 0.08], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.24, 95% CI 2-sided [-1.70 to -0.78], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.00, 95% CI 2-sided [-1.47 to -0.54], Standard Error of Mean 0.23
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.62, 95% CI 2-sided [-1.08 to -0.16], Standard Error of Mean 0.24
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.62, 95% CI 2-sided [-1.08 to -0.16], Standard Error of Mean 0.24
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.101, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.39, 95% CI 2-sided [-0.85 to 0.08], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.31, 95% CI 2-sided [-1.79 to -0.83], Standard Error of Mean 0.24
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.15, 95% CI 2-sided [-1.63 to -0.67], Standard Error of Mean 0.25
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.72, 95% CI 2-sided [-1.21 to -0.24], Standard Error of Mean 0.25
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.59, 95% CI 2-sided [-1.08 to -0.11], Standard Error of Mean 0.25
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.082, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.43, 95% CI 2-sided [-0.91 to 0.06], Standard Error of Mean 0.25

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Change at Week 2 | -1.60 (2.12) | -2.34 (2.37) | -2.33 (2.50) | -2.52 (2.40)
  Change at Week 4 | -1.84 (2.25) | -3.09 (2.49) | -3.05 (2.78) | -2.58 (2.37)
  Change at Week 8 | -1.92 (2.29) | -3.13 (2.57) | -3.10 (2.76) | -2.56 (2.34)
  Change at Week 12 | -2.03 (2.52) | -3.36 (2.58) | -3.36 (2.85) | -2.70 (2.49)
  Change at Week 16 | -2.08 (2.55) | -3.38 (2.57) | -3.30 (2.87) | -2.60 (2.59)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.70, 95% CI 2-sided [-1.12 to -0.27], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.66, 95% CI 2-sided [-1.09 to -0.23], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.82, 95% CI 2-sided [-1.25 to -0.39], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.572, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.12, 95% CI 2-sided [-0.31 to 0.55], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.467, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.16, 95% CI 2-sided [-0.27 to 0.59], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.27, 95% CI 2-sided [-1.73 to -0.82], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.15, 95% CI 2-sided [-1.61 to -0.70], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.70, 95% CI 2-sided [-1.16 to -0.24], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.57, 95% CI 2-sided [-1.03 to -0.11], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.053, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.45, 95% CI 2-sided [-0.91 to 0.01], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.21, 95% CI 2-sided [-1.66 to -0.75], Standard Error of Mean 0.23
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.11, 95% CI 2-sided [-1.56 to -0.65], Standard Error of Mean 0.23
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.61, 95% CI 2-sided [-1.07 to -0.16], Standard Error of Mean 0.23
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.59, 95% CI 2-sided [-1.05 to -0.14], Standard Error of Mean 0.23
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.035, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.49, 95% CI 2-sided [-0.95 to -0.03], Standard Error of Mean 0.23
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.32, 95% CI 2-sided [-1.79 to -0.85], Standard Error of Mean 0.24
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.24, 95% CI 2-sided [-1.71 to -0.76], Standard Error of Mean 0.24
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.64, 95% CI 2-sided [-1.11 to -0.16], Standard Error of Mean 0.24
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.68, 95% CI 2-sided [-1.16 to -0.21], Standard Error of Mean 0.24
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.013, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.60, 95% CI 2-sided [-1.07 to -0.12], Standard Error of Mean 0.24
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.29, 95% CI 2-sided [-1.76 to -0.81], Standard Error of Mean 0.24
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -1.11, 95% CI 2-sided [-1.58 to -0.63], Standard Error of Mean 0.24
Statistical Analysis 23: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.050, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.47, 95% CI 2-sided [-0.95 to -0.00], Standard Error of Mean 0.24
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.81, 95% CI 2-sided [-1.29 to -0.34], Standard Error of Mean 0.24
Statistical Analysis 25: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.63, 95% CI 2-sided [-1.11 to -0.16], Standard Error of Mean 0.24

8. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8 and 12: Baseline Observation Carried Forward (BOCF)
Description: Patient global assessment of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1=very good (no symptom and limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Change at Week 2 | -0.52 (0.87) | -0.65 (0.90) | -0.60 (0.99) | -0.88 (0.85)
  Change at Week 4 | -0.55 (0.84) | -0.90 (0.98) | -0.93 (1.03) | -0.85 (0.83)
  Change at Week 8 | -0.51 (0.84) | -0.91 (0.91) | -0.85 (1.01) | -0.71 (0.86)
  Change at Week 12 | -0.55 (0.85) | -0.85 (0.93) | -0.80 (0.93) | -0.65 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.20, 95% CI 2-sided [-0.35 to -0.04], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.113, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.12, 95% CI 2-sided [-0.28 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.34, 95% CI 2-sided [-0.49 to -0.18], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.076, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.14, 95% CI 2-sided [-0.01 to 0.29], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.21, 95% CI 2-sided [0.06 to 0.37], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.40, 95% CI 2-sided [-0.56 to -0.24], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.42, 95% CI 2-sided [-0.58 to -0.26], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.27, 95% CI 2-sided [-0.43 to -0.11], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.102, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.13, 95% CI 2-sided [-0.29 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.066, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.15, 95% CI 2-sided [-0.31 to 0.01], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.44, 95% CI 2-sided [-0.60 to -0.28], Standard Error of Mean 0.08
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.37, 95% CI 2-sided [-0.53 to -0.21], Standard Error of Mean 0.08
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.18, 95% CI 2-sided [-0.34 to -0.02], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.26, 95% CI 2-sided [-0.42 to -0.10], Standard Error of Mean 0.08
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.33, 95% CI 2-sided [-0.49 to -0.17], Standard Error of Mean 0.08
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.27, 95% CI 2-sided [-0.43 to -0.11], Standard Error of Mean 0.08
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.328, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08], Standard Error of Mean 0.08
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.09], Standard Error of Mean 0.08
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.022, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.08

9. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 8
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Change at Week 2 | -0.52 (0.87) | -0.65 (0.90) | -0.60 (0.99) | -0.88 (0.85)
  Change at Week 4 | -0.55 (0.88) | -0.91 (0.99) | -0.92 (1.05) | -0.86 (0.85)
  Change at Week 8 | -0.52 (0.90) | -0.92 (0.92) | -0.88 (1.06) | -0.78 (0.87)
  Change at Week 12 | -0.59 (0.94) | -0.95 (0.95) | -0.88 (1.00) | -0.78 (0.86)
  Change at Week 16 | -0.55 (0.91) | -0.90 (0.92) | -0.89 (1.06) | -0.79 (0.92)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.20, 95% CI 2-sided [-0.35 to -0.04], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.113, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.12, 95% CI 2-sided [-0.28 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.34, 95% CI 2-sided [-0.49 to -0.18], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.076, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.14, 95% CI 2-sided [-0.01 to 0.29], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = 0.21, 95% CI 2-sided [0.06 to 0.37], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.57 to -0.26], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.57 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.29, 95% CI 2-sided [-0.45 to -0.13], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.120, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.13, 95% CI 2-sided [-0.29 to 0.03], Standard Error of Mean 0.08
Statistical Analysis 10: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.126, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.13, 95% CI 2-sided [-0.29 to 0.04], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.46, 95% CI 2-sided [-0.62 to -0.30], Standard Error of Mean 0.08
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.57 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 13: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.08], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.009, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.22, 95% CI 2-sided [-0.38 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 15: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.052, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.16, 95% CI 2-sided [-0.32 to 0.00], Standard Error of Mean 0.08
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.57 to -0.25], Standard Error of Mean 0.08
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.31, 95% CI 2-sided [-0.48 to -0.15], Standard Error of Mean 0.08
Statistical Analysis 18: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.051, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.16, 95% CI 2-sided [-0.33 to 0.00], Standard Error of Mean 0.08
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.08], Standard Error of Mean 0.08
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.069, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.15, 95% CI 2-sided [-0.32 to 0.01], Standard Error of Mean 0.08
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 5 mg + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.41, 95% CI 2-sided [-0.57 to -0.24], Standard Error of Mean 0.08
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 10 mg + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.37, 95% CI 2-sided [-0.53 to -0.20], Standard Error of Mean 0.08
Statistical Analysis 23: Comparison: Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.21, 95% CI 2-sided [-0.37 to -0.05], Standard Error of Mean 0.08
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.20, 95% CI 2-sided [-0.36 to -0.03], Standard Error of Mean 0.08
Statistical Analysis 25: Comparison: Tanezumab 10 mg + Placebo vs Naproxen + Placebo; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value was based on pairwise comparisons; LS Mean Difference = -0.16, 95% CI 2-sided [-0.32 to 0.01], Standard Error of Mean 0.08

10. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: Participants were considered as OMERACT-OARSI responder: if the improvement from baseline to week of interest was greater than or equal to (>=) 50 percent and >=2 units in WOMAC pain subscale or WOMAC physical function subscale score; if improvement from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [worst possible pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = worse physical function) and PGA of osteoarthritis (score: 1 [very good] to 5 [very poor], higher score = worse condition). Percentage of participants who were considered as OMERACT-OARSI responder were reported in this outcome measure.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2 | 49.8 | 59.7 | 55.3 | 68.6
  Week 4 | 45.9 | 72.5 | 63.9 | 67.1
  Week 8 | 46.9 | 72.0 | 60.6 | 64.3
  Week 12 | 42.6 | 64.5 | 59.6 | 58.9
  Week 16 | 42.6 | 64.9 | 55.8 | 53.1

11. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Response at Weeks 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: Participants were considered as OMERACT-OARSI responder: if the improvement from baseline to week of interest was >=50 percent and >=2 units in WOMAC pain subscale or WOMAC physical function subscale score; if improvement from baseline to week of interest was >=20 percent and >=1 unit in at least 2 of the following: 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [worst possible pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = worse physical function) and PGA of osteoarthritis (score: 1 [very good] to 5 [very poor], higher score = worse condition). Percentage of participants who were considered as OMERACT-OARSI responder were reported in this outcome measure.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2 | 49.8 | 59.7 | 55.3 | 68.6
  Week 4 | 48.8 | 74.4 | 65.9 | 69.6
  Week 8 | 53.1 | 74.9 | 66.8 | 69.6
  Week 12 | 53.6 | 73.5 | 69.7 | 68.1
  Week 16 | 55.0 | 74.9 | 68.8 | 64.3

12. Secondary Outcome: Percentage of Participants With at Least 30 Percent and 50 Percent Reduction From Baseline in WOMAC Pain Subscale Score at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants with at least 30 percent and 50 percent reduction in WOMAC pain subscale at specified weeks were reported in this outcome measure.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2: >=30 percent reduction | 43.1 | 50.2 | 45.2 | 56.5
  Week 2: >=50 percent reduction | 26.3 | 37.0 | 28.4 | 37.2
  Week 4: >=30 percent reduction | 46.4 | 68.7 | 58.2 | 57.0
  Week 4: >=50 percent reduction | 34.0 | 51.7 | 44.2 | 39.1
  Week 8: >=30 percent reduction | 39.7 | 68.2 | 54.8 | 57.5
  Week 8: >=50 percent reduction | 32.1 | 54.0 | 42.8 | 41.1
  Week 12: >=30 percent reduction | 40.2 | 64.0 | 56.3 | 52.7
  Week 12: >=50 percent reduction | 32.1 | 53.1 | 48.6 | 41.5
  Week 16: >=30 percent reduction | 39.2 | 62.1 | 52.9 | 51.7
  Week 16: >=50 percent reduction | 29.7 | 51.7 | 44.7 | 41.1

13. Secondary Outcome: Percentage of Participants With at Least 30 Percent and 50 Percent Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 12
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2: >=30 percent reduction | 43.1 | 50.2 | 45.2 | 56.5
  Week 2: >=50 percent reduction | 26.3 | 37.0 | 28.4 | 37.2
  Week 4: >=30 percent reduction | 49.3 | 70.1 | 59.6 | 58.5
  Week 4: >=50 percent reduction | 35.9 | 53.1 | 45.2 | 40.6
  Week 8: >=30 percent reduction | 45.5 | 70.6 | 61.5 | 60.9
  Week 8: >=50 percent reduction | 35.9 | 56.4 | 47.1 | 44.4
  Week 12: >=30 percent reduction | 48.8 | 71.6 | 65.9 | 58.0
  Week 12: >=50 percent reduction | 37.8 | 58.3 | 53.8 | 45.9
  Week 16:>=30 percent reduction | 48.8 | 71.1 | 64.4 | 58.9
  Week 16:>=50 percent reduction | 35.4 | 58.8 | 51.0 | 46.9

14. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: PGA of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded on a scale ranging from 1=very good (no symptom and limitation of normal activities), 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (very severe symptoms and inability to carry out all normal activities). Higher scores indicated worse condition. Improvement signifies a decrease of at least 2 points on the 5-point scale relative to baseline value. Percentage of participants with improvement of at least 2 points in PGA of osteoarthritis were reported.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2 | 13.4 | 14.7 | 16.8 | 23.2
  Week 4 | 12.4 | 24.2 | 26.4 | 21.7
  Week 8 | 12.4 | 26.5 | 26.9 | 15.5
  Week 12 | 12.9 | 23.2 | 22.1 | 15.0
  Week 16 | 12.4 | 21.8 | 22.6 | 19.3

15. Secondary Outcome: Percentage of Participants With at Least 2 Points Improvement in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 16: Last Observation Carried Forward (LOCF)
Description: as for outcome 14
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  Week 2 | 13.4 | 14.7 | 16.8 | 23.2
  Week 4 | 12.9 | 24.6 | 26.9 | 22.2
  Week 8 | 12.4 | 27.0 | 28.8 | 17.4
  Week 12 | 13.9 | 25.6 | 25.5 | 17.9
  Week 16 | 13.4 | 24.6 | 26.0 | 21.3

16. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline up to Week 16 in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants with cumulative reduction (as percent) (greater than 0 percent [%]; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 % and 90%; = 100 %) in WOMAC pain subscale from Baseline up to Week 16 were reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  >0% reduction | 54.1 | 71.6 | 64.9 | 67.1
  >=10% reduction | 51.2 | 69.7 | 61.5 | 61.4
  >=20% reduction | 44.5 | 66.4 | 57.2 | 55.1
  >=30% reduction | 39.2 | 62.1 | 52.9 | 51.7
  >=40% reduction | 33.5 | 56.9 | 47.6 | 43.5
  >=50% reduction | 29.7 | 51.7 | 44.7 | 41.1
  >=60% reduction | 26.8 | 44.5 | 38.9 | 32.9
  >=70% reduction | 19.6 | 38.9 | 29.3 | 23.7
  >=80% reduction | 13.4 | 23.7 | 22.6 | 19.3
  >=90% reduction | 8.6 | 13.3 | 13.9 | 9.2
  =100% reduction | 2.4 | 6.2 | 5.8 | 3.4

17. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline up to Week 16 in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as the mean of scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants with cumulative reduction (as percent) (greater than 0%; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 % and 90%; = 100 %) in WOMAC pain subscale from Baseline up to Week 16 were reported.
Time Frame: Baseline up to Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
percentage of participants
  >0% reduction | 81.3 | 89.6 | 86.5 | 85.0
  >=10% reduction | 72.7 | 83.4 | 79.8 | 75.4
  >=20% reduction | 59.3 | 78.7 | 72.6 | 65.7
  >=30% reduction | 48.8 | 71.1 | 64.4 | 58.9
  >=40% reduction | 40.7 | 64.5 | 56.3 | 50.7
  >=50% reduction | 35.4 | 58.8 | 51.0 | 46.9
  >=60% reduction | 29.2 | 49.8 | 44.2 | 37.7
  >=70% reduction | 20.6 | 42.2 | 32.2 | 26.6
  >=80% reduction | 13.9 | 25.6 | 24.5 | 21.7
  >=90% reduction | 9.1 | 14.2 | 14.9 | 10.6
  =100% reduction | 2.9 | 6.2 | 6.3 | 4.3

18. Secondary Outcome: Change From Baseline in Average Daily Pain Score in the Index Hip or Knee at Weeks 2, 4, 8, 12, and 16: Baseline Observation Carried Forward (BOCF)
Description: Participants assessed their average daily pain score in the index hip/knee using a scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicated higher pain. A weekly mean was calculated using the daily index hip/knee pain scores within each specified study week. Change from baseline was calculated using the difference between each post-baseline weekly mean and the baseline mean score.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 207 | 206 | 206 | 211
units on a scale
  Change at Week 2 | -1.11 (2.06) | -1.75 (2.20) | -1.70 (2.32) | -2.02 (2.29)
  Change at Week 4 | -1.43 (2.25) | -2.34 (2.44) | -2.46 (2.54) | -2.11 (2.37)
  Change at Week 8 | -1.39 (2.27) | -2.33 (2.47) | -2.37 (2.59) | -2.01 (2.37)
  Change at Week 12 | -1.52 (2.46) | -2.39 (2.57) | -2.36 (2.83) | -2.02 (2.54)
  Change at Week 16 | -1.60 (2.51) | -2.38 (2.68) | -2.18 (2.80) | -1.82 (2.52)

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Week 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip).The WOMAC stiffness subscale was a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in the index joint (knee or hip) during the past 48 hours. It was calculated as mean of the scores from 2 individual questions scored on NRS of 0 (no stiffness) to 10 (worst stiffness), where higher scores indicated higher stiffness. Total score range for WOMAC stiffness subscale score was 0 (no stiffness) to 10 (worst stiffness), where higher scores indicated higher stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.19 (1.88) | 7.07 (1.67) | 7.11 (1.85) | 6.96 (1.99)
  Change at Week 2 | -1.54 (2.51) | -2.52 (2.59) | -2.39 (2.77) | -2.45 (2.51)
  Change at Week 4 | -1.69 (2.58) | -3.18 (2.63) | -3.10 (2.96) | -2.51 (2.47)
  Change at Week 8 | -1.74 (2.57) | -3.31 (2.79) | -2.90 (3.09) | -2.32 (2.41)
  Change at Week 12 | -1.72 (2.69) | -3.21 (2.84) | -3.06 (3.24) | -2.41 (2.67)
  Change at Week 16 | -1.74 (2.76) | -3.17 (2.89) | -2.95 (3.27) | -2.24 (2.70)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [worst possible pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = worse physical function) and WOMAC stiffness subscale assess the amount of stiffness experienced (score: 0 [no stiffness] to 10 [worst stiffness], higher score = higher stiffness). WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 (no difficulty) to 10 (maximum difficulty), where higher scores indicated worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.21 (1.35) | 7.06 (1.38) | 7.19 (1.39) | 7.07 (1.47)
  Change at week 2 | -1.75 (2.07) | -2.50 (2.35) | -2.38 (2.48) | -2.63 (2.31)
  Change at week 4 | -1.92 (2.28) | -3.23 (2.46) | -3.11 (2.75) | -2.68 (2.27)
  Change at week 8 | -1.91 (2.32) | -3.26 (2.58) | -2.94 (2.79) | -2.52 (2.24)
  Change at week 12 | -1.85 (2.54) | -3.22 (2.67) | -3.08 (2.98) | -2.56 (2.48)
  Change at week 16 | -1.88 (2.59) | -3.17 (2.68) | -2.94 (3.01) | -2.37 (2.53)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item (Pain When Walking on Flat Surface) at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Participants answered a question: "How much pain have you had when walking on a flat surface?". Participants responded about the amount of pain they experienced when walking on a flat surface by using a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 208 | 207
units on a scale
  Baseline | 7.36 (1.60) | 7.16 (1.61) | 7.23 (1.59) | 7.22 (1.61)
  Change at Week 2 | -2.14 (2.30) | -2.64 (2.60) | -2.44 (2.75) | -3.03 (2.68)
  Change at Week 4 | -2.18 (2.46) | -3.38 (2.83) | -3.26 (2.84) | -3.05 (2.55)
  Change at Week 8 | -2.23 (2.54) | -3.29 (2.75) | -3.00 (2.84) | -2.82 (2.71)
  Change at Week 12 | -2.21 (2.76) | -3.34 (2.90) | -3.20 (3.05) | -2.80 (2.74)
  Change at Week 16 | -2.19 (2.78) | -3.22 (2.90) | -2.95 (3.10) | -2.64 (2.81)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale (Pain When Going up or Down Stairs) at Weeks 2, 4, 8, 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Participants answered a question: "How much pain have you had when going up or down the stairs?" Participants responded about the amount of pain they experienced when going up or down stairs by using a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 208 | 211 | 208 | 207
units on a scale
  Baseline | 8.33 (1.36) | 8.05 (1.50) | 8.22 (1.38) | 8.24 (1.45)
  Change at Week 2 | -1.97 (2.33) | -2.84 (2.64) | -2.64 (2.72) | -2.93 (2.60)
  Change at Week 4 | -2.19 (2.50) | -3.54 (2.77) | -3.35 (2.94) | -3.07 (2.53)
  Change at Week 8 | -2.12 (2.57) | -3.44 (2.92) | -3.30 (2.99) | -2.88 (2.52)
  Change at Week 12 | -2.05 (2.83) | -3.43 (3.03) | -3.38 (3.15) | -2.84 (2.67)
  Change at Week 16 | -2.06 (2.85) | -3.33 (3.04) | -3.11 (3.17) | -2.61 (2.87)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: The SF-36 health survey is a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional, domain 8= mental health. Total score for each of the 8 domains were scaled from 0 (minimum) to 100 (maximum), where higher score indicated a better health related quality of life.
Time Frame: Baseline, Weeks 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). BOCF method was used to impute missing values. Here, 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
units on a scale
  Change at Week 12: General Health: number analyzed (Participants) | 209 | 209 | 209 | 209
  Change at Week 12: General Health | 1.11 (11.12) | 3.51 (13.04) | 4.02 (13.89) | 3.05 (13.72)
  Change at Week 16: General Health: number analyzed (Participants) | 209 | 209 | 209 | 209
  Change at Week 16: General Health | 1.43 (10.42) | 5.02 (12.38) | 3.41 (13.01) | 3.12 (11.52)
  Change at Week 12: Physical Function: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 12: Physical Function | 9.45 (20.05) | 18.57 (23.26) | 18.40 (26.35) | 11.78 (21.57)
  Change at Week 16: Physical Function: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 16: Physical Function | 8.80 (17.69) | 17.26 (21.04) | 15.93 (24.85) | 11.22 (20.80)
  Change at Week 12: Role Physical: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 12: Role Physical | 10.62 (23.47) | 19.43 (25.69) | 16.66 (24.67) | 13.22 (23.75)
  Change at Week 16: Role Physical: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 16: Role Physical | 8.85 (22.75) | 17.95 (26.59) | 15.22 (24.95) | 11.48 (24.21)
  Change at Week 12: Bodily Pain: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 12: Bodily Pain | 11.13 (21.91) | 21.89 (23.40) | 20.40 (24.28) | 15.06 (20.71)
  Change at Week 16: Bodily Pain: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 16: Bodily Pain | 10.33 (20.62) | 19.73 (24.00) | 17.54 (24.42) | 13.95 (19.22)
  Change at Week 12:Vitality: number analyzed (Participants) | 208 | 210 | 209 | 209
  Change at Week 12:Vitality | 3.85 (14.45) | 9.05 (15.00) | 6.52 (17.53) | 4.37 (18.21)
  Change at Week 16:Vitality: number analyzed (Participants) | 208 | 210 | 209 | 209
  Change at Week 16:Vitality | 4.75 (13.97) | 9.55 (15.76) | 6.97 (17.53) | 6.79 (17.00)
  Change at Week 12: Social Function: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 12: Social Function | 4.13 (17.16) | 10.12 (22.75) | 8.07 (22.66) | 7.24 (23.78)
  Change at Week 16: Social Function: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 16: Social Function | 5.44 (17.23) | 10.00 (20.31) | 7.30 (20.23) | 7.72 (22.69)
  Change at Week 12: Role Emotional: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 12: Role Emotional | 3.47 (19.48) | 8.02 (23.00) | 8.41 (23.96) | 1.75 (28.39)
  Change at Week 16: Role Emotional: number analyzed (Participants) | 209 | 210 | 209 | 209
  Change at Week 16: Role Emotional | 3.79 (18.43) | 8.49 (22.13) | 7.93 (23.02) | 3.71 (25.24)
  Change at Week 12: Mental Health: number analyzed (Participants) | 208 | 210 | 209 | 209
  Change at Week 12: Mental Health | 1.42 (12.91) | 3.17 (13.29) | 3.33 (15.44) | 3.09 (15.88)
  Change at Week 16: Mental Health: number analyzed (Participants) | 208 | 210 | 209 | 209
  Change at Week 16: Mental Health | 1.59 (11.64) | 3.74 (12.35) | 3.52 (15.81) | 2.89 (13.60)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Aggregate Scores at Weeks 12 and 16: Baseline Observation Carried Forward (BOCF)
Description: The SF-36 health survey is a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional, domain 8= mental health. Total score for each of the 8 domains were scaled from 0 (minimum) to 100 (maximum). These 8 domains are also summarized as 2 summary scores: mental component aggregate (MCA) and physical component aggregate (PCA). Total score range for each of the 2 summary scores =0 (minimum level of functioning) to 100 (maximum level of functioning). Higher (8 domains and 2 summary) scores indicate a better health related quality of life.
Time Frame: Baseline, Weeks 12, and 16
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
units on a scale
  Change at Week 12: MCA: number analyzed (Participants) | 208 | 209 | 209 | 209
  Change at Week 12: MCA | 0.01 (0.73) | 0.10 (0.85) | 0.09 (0.90) | 0.01 (1.06)
  Change at Week 16: MCA: number analyzed (Participants) | 208 | 209 | 209 | 209
  Change at Week 16: MCA | 0.07 (0.67) | 0.16 (0.81) | 0.12 (0.87) | 0.10 (0.90)
  Change at Week 12: PCA: number analyzed (Participants) | 208 | 209 | 209 | 209
  Change at Week 12: PCA | 0.43 (0.78) | 0.83 (0.99) | 0.77 (0.95) | 0.58 (0.81)
  Change at Week 16: PCA: number analyzed (Participants) | 208 | 209 | 209 | 209
  Change at Week 16: PCA | 0.39 (0.72) | 0.76 (0.95) | 0.66 (0.94) | 0.52 (0.76)

25. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). BOCF method was used to impute missing values.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
days | NA [7.0 to 106.0] — Median was not estimable due to less than 50% of population with event to meet the threshold for Kaplan-Meier analysis. | NA [10.0 to 85.0] — Median was not estimable due to less than 50% of population with event to meet the threshold for Kaplan-Meier analysis. | NA [8.0 to 92.0] — Median was not estimable due to less than 50% of population with event to meet the threshold for Kaplan-Meier analysis. | NA [7.0 to 78.0] — Median was not estimable due to less than 50% of population with event to meet the threshold for Kaplan-Meier analysis.

26. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method.
Time Frame: Baseline up to Week 16
Population: as for outcome 25
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
days | 87.78 (2.23) | 80.12 (1.09) | 84.62 (1.37) | 72.87 (1.07)

27. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. Percentage of participants with any use of rescue medication during the specified study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). LOCF method was used to impute missing values. Here 'number analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
percentage of participants
  Week 2: number analyzed (Participants) | 203 | 207 | 206 | 208
  Week 2 | 61.6 | 63.3 | 68.9 | 46.6
  Week 4: number analyzed (Participants) | 204 | 208 | 206 | 208
  Week 4 | 52.5 | 47.1 | 45.6 | 36.5
  Week 8: number analyzed (Participants) | 205 | 208 | 206 | 209
  Week 8 | 47.8 | 38.9 | 37.9 | 35.4
  Week 12: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 12 | 42.7 | 33.2 | 33.5 | 33.5
  Week 16: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 16 | 37.4 | 33.2 | 33.5 | 30.1

28. Secondary Outcome: Duration of Rescue Medication Use
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. Number of days participants used any of the rescue medication, during the specified week were summarized.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 27
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
days
  Week 2: number analyzed (Participants) | 203 | 207 | 206 | 208
  Week 2 | 1 [0 to 7] | 2 [0 to 7] | 2 [0 to 7] | 0 [0 to 7]
  Week 4: number analyzed (Participants) | 204 | 208 | 206 | 208
  Week 4 | 1 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 8: number analyzed (Participants) | 205 | 208 | 206 | 209
  Week 8 | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 12: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 12 | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 16: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 16 | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]

29. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days per week could be taken as rescue medication. The total dosage of acetaminophen in mg used during the specified week were summarized.
Time Frame: Weeks 2, 4, 8, 12, and 16
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
mg
  Week 2: number analyzed (Participants) | 203 | 207 | 206 | 208
  Week 2 | 3967.98 (5614.49) | 3661.84 (5025.34) | 3325.24 (4143.00) | 2069.71 (3851.87)
  Week 4: number analyzed (Participants) | 204 | 208 | 206 | 208
  Week 4 | 3392.16 (5588.13) | 2442.31 (4423.97) | 2648.06 (4653.47) | 1713.94 (3652.96)
  Week 8: number analyzed (Participants) | 205 | 208 | 206 | 209
  Week 8 | 3329.27 (5733.90) | 2024.04 (4124.50) | 2274.27 (4692.11) | 1956.94 (4967.74)
  Week 12: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 12 | 3055.83 (5712.68) | 2012.02 (4261.23) | 1963.59 (4531.99) | 1851.67 (3918.89)
  Week 16: number analyzed (Participants) | 206 | 208 | 206 | 209
  Week 16 | 3155.34 (5899.37) | 1968.75 (4265.10) | 2014.56 (4631.26) | 1827.75 (4138.99)

30. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 24 that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
Participants
  AEs | 85 | 101 | 101 | 110
  SAEs | 4 | 3 | 4 | 9

31. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory values: hematology (hemoglobin; hematocrit; red blood cell count [less than {<}0.8* lower limit of normal [LLN], platelets <0.5* LLN,>1.75* upper limit of normal (ULN), white blood cell count<0.6* LLN, >1.5* ULN, liver function (total bilirubin>1.5* ULN, aspartate aminotransferase; alanine aminotransferase; gamma-glutamyltransferase, lactate dehydrogenase, alkaline phosphatase>3.0* ULN, total protein; albumin<0.8* LLN; >1.2* ULN), renal function (blood urea nitrogen; creatinine>1.3* ULN, uric acid>1.2* ULN), lipids (cholesterol, triglycerides >1.3*ULN), electrolytes (sodium<0.95* LLN, >1.05* ULN; potassium; chloride; calcium; magnesium; phosphate; bicarbonate<0.9* LLN, >1.1* ULN), chemistry (glucose <0.6*LLN, >1.5*ULN; creatine kinase >2.0*ULN), urinalysis (specific gravity <1.003, >1.030; pH<4.5, >8, glucose; protein; blood; ketones; urobilinogen; bilirubin; nitrite, esterase>=1).
Time Frame: Baseline (Day 1) up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 201 | 205 | 201 | 204
Participants | 145 | 145 | 144 | 164

32. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: All standard intervals (PR, QRS, QT, QT interval corrected for heart rate using Fridericia's formula [QTcF], QT interval corrected for heart rate using Bazett's formula [QTcB], RR intervals and heart rate) were analyzed. Participants with abnormal ECG findings reported as treatment related adverse events were presented. Relatedness to treatment was assessed by investigator.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
Participants
  QRS complex abnormal | 0 | 1 | 0 | 0
  T wave abnormal | 0 | 0 | 1 | 0
  T wave inversion | 0 | 0 | 1 | 0
  Bradycardia | 0 | 0 | 1 | 0
  Ventricular extrasystoles | 0 | 0 | 1 | 0

33. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 6, 8, 12, 16 and 24
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, where 24 items scored from 0 (normal function) to 4 (extreme abnormal function), higher score indicates higher abnormality and 13 items scored from 0 (normal function) to 2 (extreme abnormal function), higher score indicates higher abnormality. NIS possible overall score ranged from 0 (no impairment) to 122 (maximum impairment), higher scores indicated increased impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). Here 'number analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
units on a scale
  Baseline: number analyzed (Participants) | 206 | 210 | 209 | 208
  Baseline | 1.52 (3.29) | 1.38 (3.04) | 0.92 (2.64) | 1.14 (3.18)
  Change at Week 2: number analyzed (Participants) | 195 | 202 | 201 | 198
  Change at Week 2 | -0.22 (1.40) | -0.21 (1.65) | 0.00 (1.85) | -0.08 (1.60)
  Change at Week 4: number analyzed (Participants) | 177 | 193 | 194 | 188
  Change at Week 4 | -0.26 (1.87) | -0.13 (1.75) | -0.26 (2.13) | -0.18 (1.54)
  Change at Week 8: number analyzed (Participants) | 157 | 185 | 172 | 173
  Change at Week 8 | -0.31 (1.52) | -0.15 (1.66) | -0.19 (1.65) | -0.17 (1.78)
  Change at Week 12: number analyzed (Participants) | 128 | 162 | 152 | 154
  Change at Week 12 | -0.29 (1.63) | -0.32 (1.55) | 0.10 (2.64) | -0.28 (1.78)
  Change at Week 16: number analyzed (Participants) | 124 | 159 | 145 | 150
  Change at Week 16 | -0.52 (1.68) | -0.25 (1.37) | -0.13 (1.54) | -0.30 (1.80)

34. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Level
Description: Participants who developed anti-tanezumab antibodies after treatment were evaluated for the presence of anti-tanezumab neutralizing antibodies in their serum. Number of participants with positive ADA were summarized for reporting groups: Tanezumab 5 mg + Placebo and Tanezumab 10 mg + Placebo. Results with titer value >= 4.32 nanogram per milliliter of anti-tanezumab neutralizing antibodies were counted as positive.
Time Frame: Baseline, Weeks 8, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure. This outcome measure was planned not to be analyzed for reporting arms: Placebo and Naproxen + Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo
Number analyzed (Participants) | 211 | 209
Participants
  Baseline | 0 | 1
  Week 8 | 1 | 0
  Week 16 | 0 | 0
  Week 24 | 0 | 0

35. Secondary Outcome: Number of Participants With Abnormal Physical Examinations Findings
Description: Physical examination included an examination of the general appearance, skin, heart, head, eyes, ears, nose, throat, breasts, abdomen, musculoskeletal, neck, extremities, thyroid and others. Criteria for abnormal physical findings were based on investigator's discretion.
Time Frame: Baseline (Day 1)
Population: ITT analysis set included all randomized participants who received at least 1 dose of randomized IV study drug (either tanezumab or IV placebo). Here, 'number analyzed' signifies those participants who were evaluable for each specified category for each group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
Participants
  Abdomen: number analyzed (Participants) | 209 | 211 | 209 | 210
  Abdomen | 19 | 12 | 11 | 15
  Ears | 5 | 11 | 7 | 6
  Extremities: number analyzed (Participants) | 206 | 208 | 208 | 209
  Extremities | 40 | 47 | 29 | 33
  Eyes | 9 | 11 | 6 | 15
  General | 14 | 12 | 3 | 17
  Head | 6 | 3 | 5 | 8
  Heart | 7 | 6 | 5 | 8
  Lungs | 5 | 3 | 1 | 1
  Musculoskeletal: number analyzed (Participants) | 206 | 209 | 208 | 209
  Musculoskeletal | 87 | 89 | 81 | 88
  Neck | 7 | 4 | 4 | 2
  Nose | 2 | 0 | 1 | 0
  Skin: number analyzed (Participants) | 208 | 210 | 209 | 209
  Skin | 31 | 23 | 31 | 34
  Throat | 6 | 1 | 3 | 3
  Thyroid | 1 | 2 | 2 | 3

36. Secondary Outcome: Number of Participants With Adverse Events Associated With Vital Sign Measurements
Description: Vital signs included the assessment of the following: body temperature, blood pressure, heart rate and respiratory rate. Number of participants with clinically significant vital signs (based on the investigator's judgment) considered as adverse events were reported.
Time Frame: Baseline (Day 1) up to Week 24
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Number analyzed (Participants) | 209 | 211 | 209 | 211
Participants | 3 | 6 | 5 | 6

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Tanezumab 5 mg + Placebo | Tanezumab 10 mg + Placebo | Naproxen + Placebo
Serious Adverse Events (participants affected / at risk) | 4/209 | 3/211 | 4/209 | 9/211
Other Adverse Events (participants affected / at risk) | 38/209 | 69/211 | 62/209 | 58/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Tanezumab 5 mg + Placebo (N=211) | Tanezumab 10 mg + Placebo (N=209) | Naproxen + Placebo (N=211)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestine ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Tanezumab 5 mg + Placebo (N=211) | Tanezumab 10 mg + Placebo (N=209) | Naproxen + Placebo (N=211)
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 2 | 10
Fatigue (General disorders) | 1 | 1 | 6 | 0
Oedema peripheral (General disorders) | 2 | 4 | 11 | 4
Bronchitis (Infections and infestations) | 2 | 6 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 8 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 8 | 6 | 5
Urinary tract infection (Infections and infestations) | 6 | 5 | 6 | 6
Fall (Injury, poisoning and procedural complications) | 5 | 6 | 4 | 5
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 12 | 12 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 11 | 2
Burning sensation (Nervous system disorders) | 0 | 2 | 5 | 2
Dizziness (Nervous system disorders) | 3 | 2 | 5 | 3
Headache (Nervous system disorders) | 6 | 9 | 7 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 7 | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 13 | 12 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.